CLINICAL TRIAL: NCT01022502
Title: Efficacy and Safety Comparison Between Refined and Crude Indigo Naturalis Ointment in the Treatment of Psoriatic Vulgaris
Brief Title: Comparison of Refined and Crude Indigo Naturalis Ointment in Treating Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yin-ku Lin (Other)
Responsible Party: Sponsor-Investigator, Yin-ku Lin, Chief of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG280391
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis, indigo naturalis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- refined indigo naturalis ointment (Active Comparator): Refined indigo naturalis ointment was applied topically to one of 2 bilaterally symmetrical psoriatic plaque lesions of the same patient for 8 weeks, starting on the date of enrollment in the study
  Interventions: Drug: refined indigo naturalis ointment
- crude indigo naturalis ointment (Active Comparator): Crude indigo naturalis ointment was applied topically to one of 2 bilaterally symmetrical psoriatic plaque lesions of the same patient for 8 weeks, starting on the date of enrollment in the study
  Interventions: Drug: crude indigo naturalis ointment

INTERVENTIONS:
Drug: refined indigo naturalis ointment — The patients applied either refined oil extract or crude indigo naturalis ointmnet topically to each of two bilaterally symmetrical psoriatic plaque lesions for 8 weeks.
  Other Names: refined ointment
  Arms: refined indigo naturalis ointment
Drug: crude indigo naturalis ointment — The patients applied either refined oil extract or crude indigo naturalis ointmnet topically to each of two bilaterally symmetrical psoriatic plaque lesions for 8 weeks.
  Other Names: Crude ointment
  Arms: crude indigo naturalis ointment

SUMMARY:
To compare the efficacy and safety of refined indigo naturalis ointment with that of crude ointment in treating psoriasis.

DETAILED DESCRIPTION:
Our previous studies have shown that topical application of indigo naturalis significantly improves psoriatic symptoms. However, patient compliance is hindered because the preparation is unsightly and stains clothing.

To improve patient compliance, we have developed a refined formulation in which closer to natural skin tones and less prone to stain clothing. In this study, we evaluated the efficacy and safety of this refined form of oil extract ointment and compared the results with those of the original crude form of indigo naturalis ointment in treating psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients were had received a diagnosis of plaque psoriasis based on clinical assessment by two dermatologists at least a one year prior to entry into the study;
* Patients had mild to moderate plaque psoriasis with bilateral symmetric lesions; were adults aged 20 to 65 years;
* Patients were in good general health.
* Female patients of childbearing age agreed to continue using birth control measures for the duration of the study.

Exclusion Criteria:

* Patients had non-plaque (i.e., pustular, guttate, or erythrodermic) or drug-induced forms of psoriasis; total body surface involvement of more than 60%;
* Patients had a history of allergy to indigo naturalis.
* Patients were excluded if they have received systemic therapy within 4 weeks before enrollment, phototherapy within 3 weeks, or used topical psoriasis agents within 2 weeks before enrollment.
* Patients had included usage of medications that affect psoriasis during the study and unwillingness to comply with study protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, MD. PhD., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from ambulatory department of Chang Gung Memorial Hospital,in northern Taiwan between November 2009 and May 2010.
Pre-assignment Details: 41 participants recruited and screened,3 exclude ( 2 did not meet the eligibility criteria and 1 refuesed to participate).
Groups:
- All Participants: In all participants, two bilateral symmetric plaques were identified, one randomly assigned to receive refined ointment, and the other assigned to receive crude ointment. Participants were instructed to avoid cross-contamination between the two treatment sites by washing hands throughly between applications. Treatment was performed until complete clearing, up to a maxmum period of 8 weeks.
Period: Overall Study
Arm/Group | All Participants
Started | 38 (19 used the refined ointment on the right site, 19 used the crude ointment on the left site.)
Completed | 35 (3 participants withdrew at week 4,5,6,respectively.)
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — employment related reasons | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants (Refined/Crude Ointment): Two symmetrically comparable plaques on each participant were identified, one randomly assigned to receive refined ointment, and the other assigned to receive crude ointment. Photographs of the lesions were taken and lesion severity was evaluated at baseline and at week 2, 4, 6, and 8.
Arm/Group | All Participants (Refined/Crude Ointment)
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 42.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Severity Idex(PSI) at Week 8.
Description: The PSI score is comprised of the grading for scaling, erythema, and induration on a 5-point scale (where 0=absent, 1=mild, 2=moderate, 3=severe and 4=very severe) and the sum of these three items with a minimal score of 0 and a maximum of score of 12. Higher values represent a worse outcome. For expample, a highter PSI score at baseline and lower PSI score after treatment represent an improvement.
Time Frame: Baseline and Week 8
Population: Total number of participants completing the 8 week period with study intervention. The paired t-test was used to compared PSI scores between the two lesions and before treatment with those after treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Crude Indigo Naturalis Ointment: Crude indigo naturalis ointment was applied topically to one of 2 bilaterally symmetrical psoriatic plaque lesions of the same patient for 8 weeks.
- Refined Indigo Naturalis Ointment: Refined indigo naturalis ointment was applied topically to one of 2 bilaterally symmetrical psoriatic plaque lesions of the same patient for 8 weeks.
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Number analyzed (Participants) | 35 | 35
units on a scale
  Scaling | -2.0 (0.90) [-2.43 to -1.62] | -2.1 (0.87) [-2.46 to -1.65]
  Erythema | -1.7 (0.85) [-2.14 to -1.35] | -2.0 (0.80) [-2.35 to -1.59]
  Induration | -1.9 (0.82) [-2.29 to -1.60] | -2.0 (0.84) [-2.34 to -1.60]
  PSI score | -5.7 (2.34) [-6.72 to -4.71] | -6.0 (2.30) [-7.03 to -4.97]

2. Primary Outcome: Clearing Percentage of Target Plaque Area
Description: The target plaque area was rated from 0% to 100% (0%=clearance after treatment and 100%=baseline before treatment). Higher values represent a worse outcome. For expample, a lower percentage after treatment represent an improvement.
Time Frame: Baseline and Week 8
Population: Total number of participants completing the 8 week period with study intervention. The paired t-test was used to compared clearing percent of target plaque between the two lesions and before treatment with those after treatment.
Measure: Mean (95% Confidence Interval); unit: percentage of the target area
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Number analyzed (Participants) | 35 | 35
percentage of the target area | 38.85 [24.48 to 53.22] | 40.97 [22.54 to 59.40]

3. Primary Outcome: Percentage Improvement Compared to Baseline in the Target Plaque.
Description: The improvement percentage of the target plaque at the follow-up visit was calculated as: [(Area of baseline plaque*PSI of baseline plaque - Area of plaque week 8*PSI of plaque week 8)/(Area of baseline plaque*PSI of baseline plaque)]*100%. Higher values represent a better outcome. For expample, a higher percent represents an improvement.
Time Frame: Baseline and Week 8
Population: Total number of participants completing the 8 week period with study intervention. The paired t-test was used to compared percent of improvement related to baseline between the two lesions and before treatment with those after treatment.
Measure: Mean (95% Confidence Interval); unit: percent change of target plaque
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Number analyzed (Participants) | 35 | 35
percent change of target plaque | 74.80 [62.57 to 87.04] | 74.28 [59.40 to 89.16]

4. Secondary Outcome: Patients' Rating of the Overall Improvement at Week 8
Description: At week 8, patients rated an overall response to treatment (separately for each side of the body), taking into account both the extent and the degree of the disease, compared with the pretreatment condition, on a 6-point scale (0=worse,1=poor, 2=fair, 3=good, 4=excellent, 5=cleared). A score of 4 or higher represents a better outcome.
Time Frame: Baseline and Week 8
Population: Total number of participants completing the 8 week period with study intervention and who reported excellent or cleared at week 8 were used for analysis.
Measure: Number; unit: participants
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Number analyzed (Participants) | 35 | 35
participants | 21 | 23

5. Secondary Outcome: Patients Preferred Ointment Type.
Description: At the end of the trial, the patients were asked which ointment they preferred.
Time Frame: Week 8
Population: Total number of participants completing the 8 week period with study intervention.
Measure: Number; unit: participants
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Number analyzed (Participants) | 35 | 35
participants | 1 | 31

ADVERSE EVENTS:
Time Frame: Week 2,4,6 and 8(end).
Description: Adverse events were recorded at each visit and determined whether they were related to the study medication.
Groups:
- Crude Indigo Naturalis Ointment: Crude indigo naturalis ointment was prepared by mixing indigo naturalis powder with olive oil,petroleum jelly and wax.
- Refined Indigo Naturalis Ointment: Refined indigo naturalis ointment was prepared by mixing indigo naturalis powder with olive oil, filtering, then mixing with petroleum jelly and wax.
Arm/Group | Crude Indigo Naturalis Ointment | Refined Indigo Naturalis Ointment
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 3/38 | 1/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crude Indigo Naturalis Ointment (N=38) | Refined Indigo Naturalis Ointment (N=38)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — Erythematous changes occurred at the beginning of treatment and resolved after a couple of days. Patch test results revealed no allergic responses, while monitoring tests for hematology, liver and renal function showed no significant findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes